CLINICAL TRIAL: NCT01300819
Title: Multicenter, Double-blind, Placebo-controlled, Parallel-group, Phase IV Study to Assess the Effect of Rotigotine on Non-motor Symptoms in Patients With Idiopathic Parkinson's Disease
Brief Title: Placebo-controlled Study in Patients With Parkinson's Disease to Evaluate the Effect of Rotigotine on Non-motor Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP0976; 2010-021394-37 (EudraCT Number)
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Results first posted 2014-05-09 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Rotigotine; Neupro®; Non-motor symptoms
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Rotigotine (Experimental)
  Interventions: Drug: Rotigotine

INTERVENTIONS:
Other: Placebo — Placebo patches of 2, 4, 6 & 8 mg / 24 hours Daily application of Placebo patches starting at 2 mg / 24 hours (early Parkinson's Disease (PD) patients) or 4 mg / 24 hours (advanced PD patients). Dose was up-titrated in weekly increments of 2 mg / 24 hours until optimal or maximal dose was reached. Maximal dose was 8 mg / 24 hours for early PD patients and 16 mg / 24 hours for advanced PD patients.
  Optimal or maximal dose was maintained for 12 weeks followed by a de-escalation by 2 mg / 24 hours every other day.
  Arms: Placebo
Drug: Rotigotine — Rotigotine patches of 2, 4, 6, and 8 mg / 24 hours
  Once daily application of Rotigotine patches starting at 2 mg / 24 hours (early Parkinson's Disease (PD) patients) or 4 mg / 24 hours (advanced PD patients). Dose was up-titrated in weekly increments of 2 mg / 24 hours until optimal or maximal dose was reached. Maximal dose is 8 mg / 24 hours for early PD patients and 16 mg / 24 hours for advanced PD patients.
  Optimal or maximal dose was maintained for 12 weeks followed by a de-escalation by 2 mg / 24 hours every other day.
  Other Names: Neupro®
  Arms: Rotigotine

SUMMARY:
The primary objective of this study was to demonstrate that Rotigotine improves non-motor symptoms compared to Placebo in subjects with Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, ≥18 years of age
* Subject has idiopathic Parkinson's disease with at least 2 of the following cardinal signs being present: bradykinesia, resting tremor, rigidity or postural instability, and without any other known or suspected cause of Parkinsonism
* Subject has a Hoehn and Yahr stage score ≤4
* Subject has a total Non-Motor Symptoms Scale (NMSS) score ≥40
* If the subject is taking levodopa (L-DOPA), he/she must be on a stable dose of L-DOPA (in combination with benserazide or carbidopa) for at least 28 days prior to the Baseline Visit
* If the subject is receiving anticholinergics, monoamine oxidase (MAO) B inhibitors, or amantadine, he/she must have been on a stable dose for at least 28 days prior to the Baseline Visit and must be maintained on that dose for the duration of the study

Exclusion Criteria:

* Subject discontinued from previous therapy with a dopamine agonist after an adequate length of treatment, at an adequate dose, due to lack of efficacy as assessed by the investigator
* Subject is receiving therapy with 1 of the following drugs, either concurrently or within 28 days prior to the Baseline Visit: alpha-methyl dopa, metoclopramide, reserpine, neuroleptics (except specific atypical neuroleptics: olanzapine, ziprasidone, aripiprazole, clozapine, and quetiapine), monoamine oxidase-A (MAO-A) inhibitors, methylphenidate, amphetamine, or other dopamine agonists (DAs)
* Subject is receiving central nervous system (CNS) therapy (eg, sedatives, hypnotics, selective serotonin reuptake inhibitors [SSRIs], anxiolytics, or other sleep-modifying medication) unless dose has been stable daily for at least 28 days prior to the Baseline Visit and is likely to remain stable for the duration of the study
* Subject has evidence of an impulse control disorder according to the modified Minnesota Impulsive Disorders Interview at the Screening Visit (Visit 1), confirmed by a positive structured clinical interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2011-02; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (87):
- Austria (3):
  - 101, Feldbach
  - 104, Vienna
  - 107, Vienna
- Belgium (5):
  - 125, Antwerp
  - 121, Bruges
  - 122, Brussels
  - 124, Ghent
  - 131, Liège
- Bulgaria (8):
  - 44, Plovdiv
  - 52, Rousse
  - 41, Sofia
  - 45, Sofia
  - 48, Sofia
  - 49, Sofia
  - 53, Sofia
  - 42, Varna
- Czechia (5):
  - 232, Chomutov
  - 227, Litomyšl
  - 222, Ostrava-Poruba
  - 231, Pilsen
  - 233, Prague
- France (6):
  - 189, Aix-en-Provence
  - 181, Amiens
  - 186, Limoges
  - 185, Pessac
  - 184, Roanne
  - 183, Toulouse
- Germany (9):
  - 62, Berlin
  - 77, Berlin
  - 67, Bochum
  - 80, Böblingen
  - 61, Marburg
  - 79, Oldenburg
  - 114, Stuttgart
  - 65, Ulm
  - 73, Westerstede
- Hungary (7):
  - 87, Budapest
  - 88, Budapest
  - 95, Győr
  - 89, Miskolc
  - 81, Nyíregyháza
  - 84, Pécs
  - 86, Szeged
- Italy (11):
  - 254, Arcugnano
  - 267, Chieti Scalo
  - 270, Napoli
  - 266, Perugia
  - 264, Pisa
  - 257, Pozzilli
  - 262, Roma
  - 269, Treviso
  - 258, Varese
  - 252, Venezia
  - 255, Verona
- Romania (10):
  - 207, Brasov
  - 201, Bucharest
  - 213, Bucharest
  - 203, Clluj-Napoca
  - 211, Cluj-Napoca
  - 208, Sibiu
  - 217, Sibiu
  - 212, Târgu Mureş
  - 204, Timișoara
  - 209, Timișoara
- Slovakia (9):
  - 245, Banská Bystrica
  - 247, Banská Bystrica
  - 240, Bratislava
  - 242, Bratislava
  - 243, Bratislava
  - 249, Dolný Kubín
  - 250, Krompachy
  - 244, Lučenec
  - 248, Žilina
- Spain (10):
  - 157, Alicante
  - 142, Barcelona
  - 146, Barcelona
  - 143, Madrid
  - 145, Madrid
  - 147, Madrid
  - 148, Madrid
  - 158, Oviedo
  - 141, Sant Cugat (Barcelona)
  - 152, Santiago de Compostela
- Switzerland (4):
  - 24, Lugano
  - 21, Sankt Gallen
  - 26, Sargans
  - 22, Zurich

REFERENCES:
- [Derived] Antonini A, Bauer L, Dohin E, Oertel WH, Rascol O, Reichmann H, Schmid M, Singh P, Tolosa E, Chaudhuri KR. Effects of rotigotine transdermal patch in patients with Parkinson's disease presenting with non-motor symptoms - results of a double-blind, randomized, placebo-controlled trial. Eur J Neurol. 2015 Oct;22(10):1400-7. doi: 10.1111/ene.12757. Epub 2015 Jun 22. PMID 26095948
- See also: FDA safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 71 sites spread across 12 countries, with 349 subjects randomized. The study duration per subject was up to 29 weeks.
  The Participant Flow consists of patients in the Enrolled Set (ES). The Enrolled Set (ES) includes all subjects who signed the Informed Consent Form.
Pre-assignment Details: Eligibility was assessed during the Screening Period, which lasted up to 4 weeks prior to the Baseline Visit. Eligible subjects returned for a Baseline Visit, during which all Baseline assessments were performed and then the subject was randomized to either Rotigotine or Placebo.
Groups:
- Placebo: Placebo : Placebo patches of 2, 4, 6 & 8 mg / 24 hours Daily application of Placebo patches starting at 2 mg / 24 hours (early Parkinson's Disease (PD) patients) or 4 mg / 24 hours (advanced PD patients). Dose will be up-titrated in weekly increments of 2 mg / 24 hours until optimal or maximal dose is reached. Maximal dose is 8 mg / 24 hours for early PD patients and 16 mg / 24 hours for advanced PD patients.
  Optimal or maximal dose will be maintained for 12 weeks followed by a de-escalation by 2 mg / 24 hours every other day.
- Rotigotine: Rotigotine : Rotigotine patches of 2, 4, 6, and 8 mg / 24 hours
  Once daily application of Rotigotine patches starting at 2 mg / 24 hours (early Parkinson's Disease (PD) patients) or 4 mg / 24 hours (advanced PD patients). Dose will be up-titrated in weekly increments of 2 mg / 24 hours until optimal or maximal dose is reached. Maximal dose is 8 mg / 24 hours for early PD patients and 16 mg / 24 hours for advanced PD patients.
  Optimal or maximal dose will be maintained for 12 weeks followed by a de-escalation by 2 mg / 24 hours every other day.
Period: Overall Study
Arm/Group | Placebo | Rotigotine
Started | 125 | 224
Completed | 103 | 180
Not Completed | 22 | 44
Not completed — Adverse Event | 9 | 27
Not completed — Lack of Efficacy | 2 | 1
Not completed — Withdrawal by Subject | 10 | 12
Not completed — Patient was 1 month late for Visit 10 | 0 | 1
Not completed — Refusal to down titrate study drug | 0 | 1
Not completed — Administrative reason | 0 | 1
Not completed — Safety follow up not done by mistake | 0 | 1
Not completed — Follow up call was not done | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented by the Randomized Set (RS), which is defined as all subjects that signed informed consent and were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rotigotine | Total
Number analyzed (Participants) | 125 | 224 | 349
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (9.8) | 68.0 (9.4) | 67.5 (9.6)
Age, Customized [Number; unit: participants]
  < 65 years | 51 | 74 | 125
  >= 65 years | 74 | 150 | 224
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 95 | 153
  Male | 67 | 129 | 196
Region of Enrollment [Number; unit: participants]
  France | 3 | 6 | 9
  Hungary | 8 | 11 | 19
  Czech Republic | 8 | 13 | 21
  Slovakia | 15 | 28 | 43
  Spain | 12 | 23 | 35
  Belgium | 4 | 9 | 13
  Romania | 18 | 36 | 54
  Austria | 2 | 1 | 3
  Bulgaria | 30 | 51 | 81
  Germany | 15 | 24 | 39
  Switzerland | 1 | 3 | 4
  Italy | 9 | 19 | 28
Weight [Mean (Standard Deviation); unit: kilogram] | 77.52 (14.90) | 76.97 (13.66) | 77.16 (14.10)
Height [Mean (Standard Deviation); unit: centimeter] | 167.42 (10.17) | 168.54 (8.56) | 168.14 (9.17)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter] | 27.593 (4.505) | 27.047 (4.348) | 27.243 (4.406)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to the End of Maintenance in Total Nonmotor Symptoms Scale (NMSS) Score
Description: The Nonmotor Symptoms Scale (NMSS) is a validated tool for rating frequency and severity of nonmotor symptoms in Parkinson's Disease (PD). The severity and frequency of the subject's nonmotor symptoms is assessed by the investigator in the following 9 domain categories: cardiovascular, including falls; sleep/fatigue; mood/cognition; perceptual problems/hallucinations; attention/memory; gastrointestinal tract; urinary; sexual function; miscellaneous. Severity and frequency are rated using a 4-point scale ranging from 0 (none) to 3 (severe; major source of distress or disturbance to subject) for severity and from 1 (rarely) to 4 (very frequent [daily or all the time]) for frequency. The total NMSS score ranges from 0 to 350. A negative change from Baseline to end of Maintenance indicates an improvement in NMSS.
Time Frame: From Baseline (Day 1) to end of 12-week Maintenance (Day 84)
Population: This analysis was performed according to the Full Analysis Set (FAS), which is defined as all treated subjects with a baseline and post-baseline NMSS measure, and follows the intention-to-treat principle.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 120 | 207
scores on a scale | -19.1 (24.2) | -23.1 (23.4)
Statistical Analysis 1: Comparison: Placebo vs Rotigotine; Null hypothesis: mean change in the total Nonmotor Symptoms Scale (NMSS) score is the same for rotigotine- and placebo-treated group; Test type: Superiority or Other; p = 0.147, ANCOVA — Two-sided p-value is presented. No multiplicity adjustment is performed; Analysing was performed with ANCOVA model, adjusted for several terms; Mean Difference (Final Values) = -3.58, 95% CI 2-sided [-8.43 to 1.26]

2. Secondary Outcome: Change From Baseline to the End of Maintenance in Total Unified Parkinson's Disease Rating Scale (UPDRS) Part III Score
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) Part III is a scale for the assessment of function in Parkinson's Disease. UPDRS Part III measures Motor Function. It consists of 14 items with 27 questions, each ranging from 0 to 4. The sum score for the UPDRS Part III ranges from 0 to 108. A higher score indicates greater disability. A negative change from Baseline to end of Maintenance score indicates improvement.
Time Frame: From Baseline (Day 1) to end of 12-week Maintenance (Day 84)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 120 | 206
scores on a scale | -3.6 (8.3) | -5.7 (8.0)
Statistical Analysis 1: Comparison: Placebo vs Rotigotine; Test type: Superiority or Other; p = 0.002, ANCOVA — Two-sided p-value is presented. No multiplicity adjustment is performed; Analysis was performed with ANCOVA model, adjusted for several terms; Mean Difference (Final Values) = -2.60, 95% CI 2-sided [-4.27 to -0.92]

3. Secondary Outcome: Change From Baseline to the End of Maintenance in Health-related Quality of Life (HRQL) Measured by a 39-item Parkinson's Disease Questionnaire (PDQ-39)
Description: Parkinson's Disease Questionnaire - 39 (PDQ-39) is a self-administered questionnaire. It comprises of 39 questions, relating to eight key areas of health and daily activities, including both Motor and Non-motor symptoms. It is scored on a scale of zero to 100, with lower scores indicating better health and high scores more severe symptoms in change from Baseline to end of Maintenance.
Time Frame: From Baseline (Day 1) to end of 12-week Maintenance (Day 84)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 116 | 204
scores on a scale | -2.6 (12.5) | -5.9 (10.8)
Statistical Analysis 1: Comparison: Placebo vs Rotigotine; Test type: Superiority or Other; p = 0.024, ANCOVA — Two-sided p-values are presented; Testing was performed using an ANCOVA model, adjusted for several terms; Mean Difference (Final Values) = -2.79, 95% CI 2-sided [-5.21 to -0.37]

4. Secondary Outcome: Change From Baseline to the End of Maintenance in the Nonmotor Symptoms Scale Score: Subdomain Cardiovascular
Description: The Nonmotor Symptoms Scale (NMSS) is a validated tool for rating frequency and severity of nonmotor symptoms in Parkinson's Disease (PD). The severity and frequency of the subject's nonmotor symptoms is assessed by the investigator in 9 different domains. Severity (ranges: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe) and frequency (ranges: 1 = Rarely (<1/wk), 2 = Often (1/wk), 3 = Frequent (several times per week), 4 = Very Frequent (daily or all the time) are rated using a 4-point scale.
  The final score is derived from multiplying the severity score and the frequency score.
  A negative change from Baseline to end of Maintenance indicates an improvement in NMSS.
  The possible min/max final scores per subdomain are calculated as follows:
  Range of final score per subdomain: 0 - 12 per question multiplied by the number of questions per subdomain:
  Subdomain Cardiovascular (2 questions): range 0 - 24
Time Frame: From Baseline (Day 1) to end of 12-week Maintenance (Day 84)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 120 | 207
scores on a scale | -1.2 (2.8) | -1.1 (3.2)
Statistical Analysis 1: Comparison: Placebo vs Rotigotine; Test type: Superiority or Other; p = 0.773, ANCOVA — Two-sided p-value is presented. No multiplicity adjustment is performed; Analysis was performed with ANCOVA model, adjusted for several terms; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.67 to 0.50]

5. Secondary Outcome: Change From Baseline to the End of Maintenance in the Nonmotor Symptoms Scale Score: Subdomain Sleep/Fatigue
Description: The Nonmotor Symptoms Scale (NMSS) is a validated tool for rating frequency and severity of nonmotor symptoms in Parkinson's Disease (PD). The severity and frequency of the subject's nonmotor symptoms is assessed by the investigator in 9 different domains. Severity (ranges: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe) and frequency (ranges: 1 = Rarely (<1/wk), 2 = Often (1/wk), 3 = Frequent (several times per week), 4 = Very Frequent (daily or all the time) are rated using a 4-point scale.
  The final score is derived from multiplying the severity score and the frequency score.
  A negative change from Baseline to end of Maintenance indicates an improvement in NMSS.
  The possible min/max final scores per subdomain are calculated as follows:
  Range of final score per subdomain: 0 - 12 per question multiplied by the number of questions per subdomain:
  Subdomain Sleep/Fatigue (4 questions): range 0-48
Time Frame: From Baseline (Day 1) to end of 12-week Maintenance (Day 84)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 120 | 207
scores on a scale | -3.9 (5.9) | -5.4 (7.8)
Statistical Analysis 1: Comparison: Placebo vs Rotigotine; Test type: Superiority or Other; p = 0.122, ANCOVA — Two-sided p-value is presented. No multiplicity adjustment is performed; Analysis was performed with ANCOVA model, adjusted for several terms; Mean Difference (Final Values) = -1.06, 95% CI 2-sided [-2.41 to 0.29]

6. Secondary Outcome: Change From Baseline to the End of Maintenance in the Nonmotor Symptoms Scale Score: Subdomain Mood/Cognition
Description: The Nonmotor Symptoms Scale (NMSS) is a validated tool for rating frequency and severity of nonmotor symptoms in Parkinson's Disease (PD). The severity and frequency of the subject's nonmotor symptoms is assessed by the investigator in 9 different domains. Severity (ranges: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe) and frequency (ranges: 1 = Rarely (<1/wk), 2 = Often (1/wk), 3 = Frequent (several times per week), 4 = Very Frequent (daily or all the time) are rated using a 4-point scale.
  The final score is derived from multiplying the severity score and the frequency score.
  A negative change from Baseline to end of Maintenance indicates an improvement in NMSS.
  The possible min/max final scores per subdomain are calculated as follows:
  Range of final score per subdomain: 0 - 12 per question multiplied by the number of questions per subdomain:
  Subdomain Mood/Cognition (6 questions): range 0 - 72
Time Frame: From Baseline (Day 1) to end of 12-week Maintenance (Day 84)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 120 | 207
scores on a scale | -5.1 (10.0) | -6.6 (11.0)
Statistical Analysis 1: Comparison: Placebo vs Rotigotine; Test type: Superiority or Other; p = 0.047, ANCOVA — Two-sided p-value is presented. No multiplicity adjustment is performed; Analysis was performed with ANCOVA model, adjusted for several terms; Mean Difference (Final Values) = -1.81, 95% CI 2-sided [-3.59 to -0.02]

7. Secondary Outcome: Change From Baseline to the End of Maintenance in the Nonmotor Symptoms Scale Score: Subdomain Perception/Hallucinations
Description: The Nonmotor Symptoms Scale (NMSS) is a validated tool for rating frequency and severity of nonmotor symptoms in Parkinson's Disease (PD). The severity and frequency of the subject's nonmotor symptoms is assessed by the investigator in 9 different domains. Severity (ranges: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe) and frequency (ranges: 1 = Rarely (<1/wk), 2 = Often (1/wk), 3 = Frequent (several times per week), 4 = Very Frequent (daily or all the time) are rated using a 4-point scale.
  The final score is derived from multiplying the severity score and the frequency score.
  A negative change from Baseline to end of Maintenance indicates an improvement in NMSS.
  The possible min/max final scores per subdomain are calculated as follows:
  Range of final score per subdomain: 0 - 12 per question multiplied by the number of questions per subdomain:
  Subdomain Perception/Hallucinations (3 questions): range 0 - 36
Time Frame: From Baseline (Day 1) to end of 12-week Maintenance (Day 84)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 120 | 207
scores on a scale | -0.2 (1.8) | -0.2 (1.6)
Statistical Analysis 1: Comparison: Placebo vs Rotigotine; Test type: Superiority or Other; p = 0.601, ANCOVA — Two-sided p-value is presented. No multiplicity adjustment is performed; Analysis was performed with ANCOVA model, adjusted for several terms; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.22 to 0.37]

8. Secondary Outcome: Change From Baseline to the End of Maintenance in the Nonmotor Symptoms Scale Score: Subdomain Attention/Memory,
Description: The Nonmotor Symptoms Scale (NMSS) is a validated tool for rating frequency and severity of nonmotor symptoms in Parkinson's Disease (PD). The severity and frequency of the subject's nonmotor symptoms is assessed by the investigator in 9 different domains. Severity (ranges: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe) and frequency (ranges: 1 = Rarely (<1/wk), 2 = Often (1/wk), 3 = Frequent (several times per week), 4 = Very Frequent (daily or all the time) are rated using a 4-point scale.
  The final score is derived from multiplying the severity score and the frequency score.
  A negative change from Baseline to end of Maintenance indicates an improvement in NMSS.
  The possible min/max final scores per subdomain are calculated as follows:
  Range of final score per subdomain: 0 - 12 per question multiplied by the number of questions per subdomain:
  Subdomain Attention/Memory (3 questions): range 0 - 36
Time Frame: From Baseline (Day 1) to end of 12-week Maintenance (Day 84)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 120 | 207
scores on a scale | -1.3 (4.8) | -1.5 (4.7)
Statistical Analysis 1: Comparison: Placebo vs Rotigotine; Test type: Superiority or Other; p = 0.997, ANCOVA — Two-sided p-value is presented. No multiplicity adjustment is performed; Analysis was performed with ANCOVA model, adjusted for several terms; Mean Difference (Final Values) = 0, 95% CI 2-sided [-0.99 to 0.99]

9. Secondary Outcome: Change From Baseline to the End of Maintenance in the Nonmotor Symptoms Scale Score: Subdomain Gastrointestinal Tract
Description: The Nonmotor Symptoms Scale (NMSS) is a validated tool for rating frequency and severity of nonmotor symptoms in Parkinson's Disease (PD). The severity and frequency of the subject's nonmotor symptoms is assessed by the investigator in 9 different domains. Severity (ranges: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe) and frequency (ranges: 1 = Rarely (<1/wk), 2 = Often (1/wk), 3 = Frequent (several times per week), 4 = Very Frequent (daily or all the time) are rated using a 4-point scale.
  The final score is derived from multiplying the severity score and the frequency score.
  A negative change from Baseline to end of Maintenance indicates an improvement in NMSS.
  The possible min/max final scores per subdomain are calculated as follows:
  Range of final score per subdomain: 0 - 12 per question multiplied by the number of questions per subdomain:
  Subdomain Gastrointestinal tract (3 questions): range 0 - 36
Time Frame: From Baseline (Day 1) to end of 12-week Maintenance (Day 84)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 120 | 207
scores on a scale | -1.4 (3.4) | -1.6 (3.5)
Statistical Analysis 1: Comparison: Placebo vs Rotigotine; Test type: Superiority or Other; p = 0.584, ANCOVA — Two-sided p-value is presented. No multiplicity adjustment is performed; Analysis was performed with ANCOVA model, adjusted for several terms; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.87 to 0.49]

10. Secondary Outcome: Change From Baseline to the End of Maintenance in the Nonmotor Symptoms Scale Score: Subdomain Urinary
Description: The Nonmotor Symptoms Scale (NMSS) is a validated tool for rating frequency and severity of nonmotor symptoms in Parkinson's Disease (PD). The severity and frequency of the subject's nonmotor symptoms is assessed by the investigator in 9 different domains. Severity (ranges: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe) and frequency (ranges: 1 = Rarely (<1/wk), 2 = Often (1/wk), 3 = Frequent (several times per week), 4 = Very Frequent (daily or all the time) are rated using a 4-point scale.
  The final score is derived from multiplying the severity score and the frequency score.
  A negative change from Baseline to end of Maintenance indicates an improvement in NMSS.
  The possible min/max final scores per subdomain are calculated as follows:
  Range of final score per subdomain: 0 - 12 per question multiplied by the number of questions per subdomain:
  Subdomain Urinary (3 questions): range 0 - 36
Time Frame: From Baseline (Day 1) to end of 12-week Maintenance (Day 84)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 120 | 207
scores on a scale | -2.7 (6.6) | -2.4 (6.0)
Statistical Analysis 1: Comparison: Placebo vs Rotigotine; Test type: Superiority or Other; p = 0.536, ANCOVA — Two-sided p-value is presented. No multiplicity adjustment is performed; Analysis was performed with ANCOVA model, adjusted for several terms; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [-0.84 to 1.60]

11. Secondary Outcome: Change From Baseline to the End of Maintenance in the Nonmotor Symptoms Scale Score: Subdomain Sexual Function
Description: The Nonmotor Symptoms Scale (NMSS) is a validated tool for rating frequency and severity of nonmotor symptoms in Parkinson's Disease (PD). The severity and frequency of the subject's nonmotor symptoms is assessed by the investigator in 9 different domains. Severity (ranges: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe) and frequency (ranges: 1 = Rarely (<1/wk), 2 = Often (1/wk), 3 = Frequent (several times per week), 4 = Very Frequent (daily or all the time) are rated using a 4-point scale.
  The final score is derived from multiplying the severity score and the frequency score.
  A negative change from Baseline to end of Maintenance indicates an improvement in NMSS.
  The possible min/max final scores per subdomain are calculated as follows:
  Range of final score per subdomain: 0 - 12 per question multiplied by the number of questions per subdomain:
  Subdomain Sexual function (2 questions): range 0 - 24
Time Frame: From Baseline (Day 1) to end of 12-week Maintenance (Day 84)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 120 | 207
scores on a scale | -1.2 (4.2) | -1.1 (4.3)
Statistical Analysis 1: Comparison: Placebo vs Rotigotine; Test type: Superiority or Other; p = 0.889, ANCOVA — Two-sided p-value is presented. No multiplicity adjustment is performed; Analysis was performed with ANCOVA model, adjusted for several terms; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.81 to 0.94]

12. Secondary Outcome: Change From Baseline to the End of Maintenance in the Nonmotor Symptoms Scale Score: Subdomain Miscellaneous
Description: The Nonmotor Symptoms Scale (NMSS) is a validated tool for rating frequency and severity of nonmotor symptoms in Parkinson's Disease (PD). The severity and frequency of the subject's nonmotor symptoms is assessed by the investigator in 9 different domains. Severity (ranges: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe) and frequency (ranges: 1 = Rarely (<1/wk), 2 = Often (1/wk), 3 = Frequent (several times per week), 4 = Very Frequent (daily or all the time) are rated using a 4-point scale.
  The final score is derived from multiplying the severity score and the frequency score.
  A negative change from Baseline to end of Maintenance indicates an improvement in NMSS.
  The possible min/max final scores per subdomain are calculated as follows:
  Range of final score per subdomain: 0 - 12 per question multiplied by the number of questions per subdomain:
  Subdomain Miscellaneous (4 questions): range 0 - 48
Time Frame: From Baseline (Day 1) to end of 12-week Maintenance (Day 84)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 120 | 207
scores on a scale | -2.2 (4.4) | -3.2 (5.7)
Statistical Analysis 1: Comparison: Placebo vs Rotigotine; Test type: Superiority or Other; p = 0.043, ANCOVA — Two-sided p-value is presented. No multiplicity adjustment is performed; Analysis was performed with ANCOVA model, adjusted for several terms; Mean Difference (Final Values) = -1.04, 95% CI 2-sided [-2.06 to -0.03]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected during 16 weeks (from Baseline to Safety Follow up Visit).
Description: The Analysis Population refers to the Safety Set (SS). The SS consists of all randomized subjects receiving at least 1 dose of Investigational Medicinal Product (IMP).
Arm/Group | Placebo | Rotigotine
Serious Adverse Events (participants affected / at risk) | 4/125 | 8/223
Other Adverse Events (participants affected / at risk) | 21/125 | 66/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=125) | Rotigotine (N=223)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Acute cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Tachycardia paroxysmal (Cardiac disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic coma (Nervous system disorders) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Artrial Fibrillation + Chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Worsening of Parkinson's Disease (Nervous system disorders) | 0 (0) | 1 (1)
Exacerbation of chronic left sided heart insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=125) | Rotigotine (N=223)
Nausea (Gastrointestinal disorders) | 7 (8) | 27 (30)
Application site pruritus (General disorders) | 2 (3) | 15 (16)
Fatigue (General disorders) | 7 (8) | 9 (10)
Somnolence (Nervous system disorders) | 7 (8) | 18 (21)
Dizziness (Nervous system disorders) | 9 (9) | 15 (15)
Headache (Nervous system disorders) | 5 (5) | 12 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days